CLINICAL TRIAL: NCT00817245
Title: Effect of Helicobacter Pylori Treatment on Remission of Idiopathic Central Serous Chorioretinopathy (ICSCR)
Brief Title: Effect of Helicobacter Pylori Treatment on Idiopathic Central Serous Chorioretinopathy (ICSCR)
Acronym: ICSCR
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Tabriz University (Other)
Responsible Party: Alireza Javadzadeh, Tabriz University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 86-47
Record Dates: First submitted 2009-01-01; First posted 2009-01-06 (Estimated); Last update posted 2009-01-06 (Estimated); Status verified 2009-01

CONDITIONS: Central Serous Chorioretinopathy
Keywords: CSR; Helicobacter pylori
MeSH Terms: conditions — Central Serous Chorioretinopathy | interventions — Omeprazole; Amoxicillin; Metronidazole

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Oral Amoxicillin Capsule Metronidazole Tablet Omeprazole Capsule
  Interventions: Drug: omeprazole, Amoxicillin, metronidazole
- 2 (No Intervention): No medical treatment

INTERVENTIONS:
Drug: omeprazole, Amoxicillin, metronidazole — we will evaluate the effect of medication(anti h.pylori) on the remission of ICSCR
  Other Names: treatment of Central serous chorioretinopathy
  Arms: 1

SUMMARY:
Etiology of ICSCR is not known however recent studies regard the role of immunologic and infectious processes in the pathogenesis of ICSCR.one of these hypothesis is the role of helicobacter pylori in the pathogenesis of ICSCR so perhaps treatment of h pylori have positive effect on the remission of ICSCR.

DETAILED DESCRIPTION:
we will choose 50 cases of patients with ICSCR who are infected with h.pylori.25 cases will receive anti h.pylori regiment and 25 cases as controls will receive no medication.then we will compare the time of submacular fluid resorption and macular thickness and visual acuity among these two groups.

ELIGIBILITY:
Inclusion Criteria:

* the persons who are infected with helicobacter pylori and have ICSCR

Exclusion Criteria:

* history of previous eye surgery ,to have indication of laser therapy,corticosteroid therapy,pregnancy,

Ages: 28 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2008-03; Primary Completion 2008-10 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Subretinal fluid level

SECONDARY OUTCOMES:
time of sub macular fluid absorption

CONTACTS AND LOCATIONS:
Overall Officials: Alireza Javadzadeh, Study Chair — Alireza Javadzadeh
Locations (1):
- Alireza JavadzadehTabriz, Tabriz, Iran

REFERENCES:
- [Derived] Lange CA, Qureshi R, Pauleikhoff L. Interventions for central serous chorioretinopathy: a network meta-analysis. Cochrane Database Syst Rev. 2025 Jun 16;6(6):CD011841. doi: 10.1002/14651858.CD011841.pub3. PMID 40522203